CLINICAL TRIAL: NCT03769610
Title: Inpatient Versus Outpatient Transcervical Foley Catheter Use for Cervical Ripening: A Randomized Controlled Trial
Brief Title: Inpatient Versus Outpatient Cervical Ripening
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: LifeBridge Health (Other)
Collaborators: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Rebecca Pierce-Williams, Resident physician, LifeBridge Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2383
Record Dates: First submitted 2017-10-12; First posted 2018-12-07 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Pregnancy Related; Labor; Induction; Cervical Ripening
Keywords: Foley; Transcervical

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned to either inpatient or outpatient cervical ripening with a Foley catheter.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inpatient Foley catheter (Active Comparator): Subjects will be admitted to a room on labor and delivery and will be monitored with the external fetal monitor (EFM) and tocometer (a device to monitor contractions). If she is contracting less than every 2 minutes, intravenous (IV) Pitocin will be started at 2 milliunits/minute and increased per hospital protocol. While on pitocin, she will remain on continuous EFM and tocometer. She will also be kept on a clear liquid diet with intravenous fluids per standard protocol. If the Foley catheter has not been expulsed in 24 hours, it will be removed. After expulsion or removal of the Foley catheter, induction may proceed as deemed clinically appropriate by the managing physician. No further cervical ripening will be performed after the Foley catheter is expulsed/removed, or after 24 hours.
  Interventions: Other: Inpatient Foley catheter
- Outpatient Foley catheter (Experimental): Subjects are asked to return to the hospital ~12 hours after placement. Subjects are to return to the hospital if they develop heavy vaginal bleeding, decreased fetal movement, rupture of membranes, or increasingly painful or frequent contractions requiring an epidural or pain relief. Once admitted, subjects will be evaluated for expulsion of the catheter. If the catheter is in place IV Pitocin will be started. If the catheter has been expulsed, the induction will proceed as deemed clinically appropriate. After 24 hours, if the Foley catheter is still in the cervix it will be removed and the induction will proceed as deemed clinically appropriate.
  Interventions: Other: Outpatient Foley catheter

INTERVENTIONS:
Other: Inpatient Foley catheter
  Arms: Inpatient Foley catheter
Other: Outpatient Foley catheter
  Arms: Outpatient Foley catheter

SUMMARY:
Induction of labor is a process of stimulating uterine contractions before the onset of labor, with a goal of achieving vaginal birth. The cervix (the lower part of the uterus that connects to the vagina) must dilate (open) in order to allow passage of the baby into the vagina and through the birth canal. A process called "cervical ripening" is often performed prior to labor induction to prepare the cervix for labor and therefore shorten the length of the labor. There are various pharmacologic and mechanical methods of cervical ripening that result in the physical softening and distensibility of the cervix. Mechanical dilation with a small balloon (i.e. a Foley catheter) placed in the cervix is one of the most commonly used, safe, inexpensive, and effective methods to achieve cervical ripening.

In most hospitals, cervical ripening is performed in the hospitals; however, some hospitals allow women to undergo cervical ripening at home with a transcervical Foley catheter. The goal of this study is to compare the use of a Foley catheter for cervical ripening in the inpatient (in-hospital) and outpatient (at home) settings. We anticipate that outpatient use will lead to a shorter amount of time that a woman spends in the hospital, decreased cost, and good patient satisfaction.

DETAILED DESCRIPTION:
From 1990 to 2010, the rates of induction of labor increased from 9.6% to 23.8%(1). Recent data from 2014 reports a rate of 23.2%(2). Labor induction may be medically indicated, in cases in which the risk of continuing pregnancy is greater than delivery, or in some cases electively after 39 weeks of gestation.

Prior to starting an induction of labor, a digital exam is performed to determine the status of the cervix in terms of its dilatation, effacement, position, softness, and fetal station. If the cervical status is considered favorable for labor, then generally oxytocin is started to induce uterine contractions. If the cervix is not considered favorable, a method of cervical ripening is employed to induce physical changes in the cervix that make it more favorable for labor.

This process involves inflammatory infiltration and release of metalloproteases that degrade collagen and result in cervical remodeling(3). The primary benefit of cervical ripening is reducing the length of labor; however, some studies have suggested that it may lower the rate of cesarean section(4,5). The Bishop score (see table 1) is used as a scoring tool to determine the status of the cervix(6). Most studies define a score of 6 or less as an unfavorable cervix, while a score of greater than 8 is favorable, and has a similar probability of vaginal delivery to spontaneous labor(7).

Commonly used methods for cervical ripening include pharmacologic forms such as synthetic prostaglandin E1 (PGE1, i.e. misoprostol) and prostaglandin E2 (PGE2, i.e. dinoprostone), or mechanical ripening with balloon (i.e. Foley) catheters.

Quality improvement, increasing efficiency, and decreasing cost continue to be challenges for individual hospitals and the entire health care system. Induction of labor, especially with an unfavorable cervix, is associated with longer lengths of stay for patients, which results in increased cost(8).

Foley catheters are a safe, inexpensive and effective option for cervical ripening. A study by Sciscione et al in 2001 compared Foley bulb use in inpatient versus outpatient settings and found the outpatient use to be as effective for cervical ripening. The primary objective of this study was to compare efficacy of these two approaches and the outcomes were similar. There were no cases of endomyometritis or chorioamnionitis(9). While they did report a shorter amount of time in the hospital with outpatient management, this was not a primary outcome of the study and they did not compare costs. Recently there has been an increased focus on the costs of medical care and patient satisfaction. Consequently, these are increasingly important outcomes that research needs to focus on. It is our hope that the findings of our study will support the use of outpatient pre-induction of labor cervical ripening and result in a more efficient use of resources and improved patient satisfaction.

The purpose of this study is to compare the use of a Foley catheter for cervical ripening in the inpatient and outpatient setting, in order to evaluate the difference in the amount of time spent on labor and delivery during induction of labor, as well as the difference in costs. An important secondary outcome we plan to evaluate as well is patient satisfaction. This will be a randomized controlled trial, with the study population being pregnant women at ≥ 37 weeks of gestation undergoing induction of labor. The projected time-frame will be from October 2016 to June 2018. The expected outcome is that outpatient cervical ripening with Foley catheter use will result in shorter lengths of stay on labor and delivery and less cost than inpatient Foley catheter use in patients undergoing induction of labor. Additionally, we anticipate greater patient satisfaction with outpatient management.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancies at least 37 weeks' gestation, undergoing induction of labor, with an unfavorable cervix, defined as a Bishop score ≤ 6
* The fetus must be in the cephalic presentation
* Indications for induction of labor include, but are not limited to, the following:

  * Elective induction of labor at 39 weeks' gestation
  * Intrauterine growth restriction
  * Chronic hypertension
  * Diabetes
  * Gestational diabetes
  * Prior stillbirth
  * Other medical indications for induction of labor, as deemed appropriate by the obstetric provider, such as Systemic Lupus Erythematosus, Cholestasis of Pregnancy etc.

Exclusion Criteria:

* Gestational hypertension
* Preeclampsia
* Non-reassuring fetal testing
* Multi-fetal gestation
* Oligohydramnios
* Fetal anomaly
* Less than 37 weeks
* Bishop score > 6
* Ruptured membranes
* Contraindication to vaginal delivery including: active Herpes lesion, HIV VL >1000 copies/mL, placenta previa, vasa previa, breech presentation, prior classical cesarean section or transfundal myomectomy
* Poor access to telephone or transportation
* Latex allergy
* Any other condition for which the managing physician or investigator deem outpatient management inappropriate.
* Currently participating in another clinical trial

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Pregnant women
Enrollment: 30 (Actual)
Dates: Start 2017-01-04 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Difference in time on labor and delivery | (approximately) 2 days
  To evaluate the difference in the amount of time a patient spends on labor and delivery during induction of labor when undergoing inpatient versus outpatient transcervical Foley catheter for induction of labor.
Difference in cost | (approximately 5 days)
  To compare the difference in cost for hospitalization in patients undergoing inpatient versus outpatient cervical ripening with a transcervical Foley catheter.

SECONDARY OUTCOMES:
Patient satisfaction | (approximately 5 days)
  Each subject is asked to complete a survey
Provider satisfaction | (approximately 3 years)
  After enrollment is completed, providers will be surveyed on their satisfaction
Length of labor induction | (approximately 3 days)
  Total length of induction, including cervical ripening
Type of delivery | (approximately 3 days)
  Vaginal delivery versus cesarean section
Maternal blood loss | (approximately 3 days)
  Total blood loss at delivery
Infection rates | (approximately 5 days)
  Maternal intrapartum and postpartum infections
Apgar scores | (approximately 10 minutes)
  Neonatal Apgar scores at 1 and 5 minutes, and 10 minutes if reported
Non-reassuring fetal heart tracings | (approximately 3 days)
  Any non-reassuring fetal monitoring during labor

OTHER OUTCOMES:
NICU admission | (approximately 5 days)
  Any neonatal ICU admissions
Neonatal fever | (approximately 5 days)
  Any neonatal fever
Total time on pitocin | (approximately 3 days)
  Time on pitocin for induction
Maximum dose of pitocin | (approximately 3 days)
  Max dose

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Thomas Jefferson University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martin JA, Hamilton BE, Osterman MJ, Curtin SC, Matthews TJ. Births: final data for 2013. Natl Vital Stat Rep. 2015 Jan 15;64(1):1-65. PMID 25603115
- [Background] Hamilton BE, Martin JA, Osterman MJ, Curtin SC, Matthews TJ. Births: Final Data for 2014. Natl Vital Stat Rep. 2015 Dec;64(12):1-64. PMID 26727629
- [Background] Smith R. Parturition. N Engl J Med. 2007 Jan 18;356(3):271-83. doi: 10.1056/NEJMra061360. No abstract available. PMID 17229954
- [Background] Thomas J, Fairclough A, Kavanagh J, Kelly AJ. Vaginal prostaglandin (PGE2 and PGF2a) for induction of labour at term. Cochrane Database Syst Rev. 2014 Jun 19;2014(6):CD003101. doi: 10.1002/14651858.CD003101.pub3. PMID 24941907
- [Background] Jozwiak M, Bloemenkamp KW, Kelly AJ, Mol BW, Irion O, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2012 Mar 14;(3):CD001233. doi: 10.1002/14651858.CD001233.pub2. PMID 22419277
- [Background] BISHOP EH. PELVIC SCORING FOR ELECTIVE INDUCTION. Obstet Gynecol. 1964 Aug;24:266-8. No abstract available. PMID 14199536
- [Background] ACOG Practice Bulletin No. 107: Induction of labor. Obstet Gynecol. 2009 Aug;114(2 Pt 1):386-397. doi: 10.1097/AOG.0b013e3181b48ef5. No abstract available. PMID 19623003
- [Background] von Gruenigen VE, Powell DM, Sorboro S, McCarroll ML, Kim U. The financial performance of labor and delivery units. Am J Obstet Gynecol. 2013 Jul;209(1):17-9. doi: 10.1016/j.ajog.2013.02.019. Epub 2013 Feb 11. PMID 23410692
- [Background] Sciscione AC, Muench M, Pollock M, Jenkins TM, Tildon-Burton J, Colmorgen GH. Transcervical Foley catheter for preinduction cervical ripening in an outpatient versus inpatient setting. Obstet Gynecol. 2001 Nov;98(5 Pt 1):751-6. doi: 10.1016/s0029-7844(01)01579-4. PMID 11704164
- [Derived] Alfirevic Z, Gyte GM, Nogueira Pileggi V, Plachcinski R, Osoti AO, Finucane EM. Home versus inpatient induction of labour for improving birth outcomes. Cochrane Database Syst Rev. 2020 Aug 27;8(8):CD007372. doi: 10.1002/14651858.CD007372.pub4. PMID 32852803